CLINICAL TRIAL: NCT01491802
Title: A 4-week Randomized, Double-blind, Crossover Study to Assess the Effect of a New LABA/LAMA Combination Versus LAMA Alone on Exertional Dyspnea, Exercise Endurance and Neuromechanical Coupling in Patients With GOLD Stage II COPD
Brief Title: Effect of a New Combination Bronchodilator on Exercise in GOLD Stage II Moderate COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Dr. Denis O'Donnell, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMED-1426-11
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-05

CONDITIONS: COPD
Keywords: COPD; Combination therapy; Anticholinergic; Beta2-agonist; Exercise; Dyspnea; Respiratory mechanics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Dyspnea | interventions — GSK573719; vilanterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LAMA alone, then LAMA/LABA combination (Experimental): Participants will first receive an inhaled long-acting muscarinic antagonist (LAMA) once daily for 4 weeks. After a 2 week washout period, they will then receive the fixed-dose combination product [LAMA plus long-acting beta2-agonist (LABA)] once daily for 4 weeks.
  Interventions: Drug: LAMA/LABA; Drug: LAMA
- LABA/LAMA combination, then LAMA alone (Experimental): Participants will first receive a long-acting muscarinic antagonist (LAMA) plus long-acting beta2-agonist (LABA) combination product once daily for 4 weeks. After a 2 week washout period, they will then receive the LAMA single product once daily for 4 weeks.
  Interventions: Drug: LAMA/LABA; Drug: LAMA

INTERVENTIONS:
Drug: LAMA/LABA — GSK573719/GW642444 inhalation powder used in the Novel Dry Powder Inhaler (DPI): a long-acting beta2-agonist (GSK642444, 25mcg) with a long-acting muscarinic antagonist (GSK573719, 125mcg) combination therapy will be taken once daily for 4 weeks.
  Other Names: GSK573719+GW642444; umeclidinium (GSK573719) / vilanterol (GW642444); Anoro ELLIPTA
Drug: LAMA — GSK573719 (125mcg) inhalation powder is a long-acting muscarinic antagonist that will be taken once daily for 4 weeks
  Other Names: umeclidinium

SUMMARY:
Preliminary information from our laboratory indicated that even patients with milder chronic obstructive pulmonary disease (COPD) can have significant physiological derangements which become more pronounced during exercise, leading to intolerable dyspnea at lower levels of ventilation than in health. This study will explore pathophysiological mechanisms of dyspnea and activity limitation in GOLD stage II COPD and will determine if there is a sound physiological rationale for the use of dual long-acting beta2-agonist (LABA)/long-acting muscarinic antagonist (LAMA) therapy (GSK573719/ GW642444 Inhalation Powder) versus LAMA alone (GSK573719) as treatment for dyspnea and exercise intolerance in this subpopulation. Objectives of this study are to determine if: 1) neuromechanical uncoupling of the respiratory system contributes to exertional dyspnea in milder COPD, and 2) treatment with LABA/LAMA improves dyspnea and exercise endurance compared with LAMA by improving neuromechanical coupling. The investigators hypothesize that: 1) dyspnea is related to excessive dynamic lung hyperinflation, tidal volume restriction and increased ratio of central respiratory neural drive to tidal volume displacement, a measure of neuromechanical uncoupling of the respiratory system, and 2) LABA/LAMA will improve dyspnea and exercise endurance, which will be explained by partial reversal of the above mechanical abnormalities. The investigators will conduct a randomized, double-blind crossover study and compare the effects of once-daily LABA/LAMA over 4-weeks with LAMA on dyspnea, exercise endurance and ventilatory mechanics in GOLD stage II COPD.

ELIGIBILITY:
Inclusion Criteria:

* Stable moderate COPD
* Post-bronchodilator FEV1/FVC<0.7 and 50%≤FEV1<80% predicted
* Baseline Dyspnea Index ≤ 9 and MRC dyspnea scale >2
* Cigarette smoking history at least 20 pack-years

Exclusion Criteria:

* Presence of a significant disease other than COPD that could contribute to dyspnea and exercise limitation
* Important contraindications to clinical exercise testing
* Use of daytime oxygen
* History of asthma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis E O'Donnell, MD, FRCPC, Principal Investigator — Queen's University and Kingston General Hospital
Locations (1):
- Respiratory Investigation Unit at Kingston General Hospital, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between March 2012 and June 2014.
Pre-assignment Details: There was run-in period of approximately 2 weeks for determination of eligibility and familiarization with all tests to be performed during subsequent treatment visits. There was a 2-week washout period between each 4-week treatment period of this crossover study.
Groups:
- LAMA, Then LAMA/LABA: Participants first received LAMA alone (umeclidinium 125 mcg) once daily for 4 weeks. After a 2 week washout period, they received the LAMA/LABA combination product (umeclidinium 125 mcg plus vilanterol 25 mcg) once daily for 4 weeks.
- LAMA/LABA, the LAMA: Participants first received the LAMA/LABA combination product (umeclidinium 125 mcg plus vilanterol 25 mcg) once daily for 4 weeks. After a 2 week washout period, they received LAMA alone (umeclidinium 125 mcg) once daily for 4 weeks.
Period: Overall Study
Arm/Group | LAMA, Then LAMA/LABA | LAMA/LABA, the LAMA
Started | 9 | 8
Completed | 8 | 6
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Randomized Subjects: All 17 randomized subjects.
Arm/Group | Randomized Subjects
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 17
FEV1 %predicted [Mean (Standard Deviation); unit: % of predicted normal] — Post-bronchodilator measurement
  % of predicted normal | 70.9 (69.4)
FEV1/FVC % ratio [Mean (Standard Deviation); unit: %] — Post-bronchodilator measurement
  % | 55.6 (7.7)
Smoking history [Mean (Standard Deviation); unit: pack-years] | 49 (20)
Baseline Dyspnea Index score [Mean (Standard Deviation); unit: units on a scale] — Scoring range for activity-related dyspnea is 0 (most severe) to 12 (none).
  units on a scale | 7.9 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Exertional Dyspnea Intensity at Isotime Exercise.
Description: Intensity of dyspnea (defined as breathing discomfort) at a standardized time (isotime) during constant work rate exercise tests as measured by the modified 10-point Borg scale. A rating of 0 represents no dyspnea up to a maximum of 10: a smaller rating is therefore an improvement. Isotime was defined as the highest exercise time in minutes completed in both post-treatment tests.
Time Frame: 4 weeks
Population: Of the 17 randomized subjects, 3 subjects were withdrawn (2 AEs, 1 withdrawn consent ) leaving 14 completed subjects for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- LAMA: GSK573719 is a long-acting muscarinic antagonist
  GSK573719: GSK573719 (125mcg) inhalation powder is a long-acting muscarinic antagonist that will be taken once daily for 4 weeks
- LABA/LAMA Combination: GSK573719/GW642444 inhalation powder used in the Novel Dry Powder Inhaler (DPI): a long-acting beta2-agonist (GSK642444, 25mcg) with a long-acting muscarinic antagonist (GSK573719, 125mcg) combination therapy.
  GSK573719/GW642444: GSK573719/GW642444 inhalation powder used in the Novel Dry Powder Inhaler (DPI): a long-acting beta2-agonist (GSK642444, 25mcg) with a long-acting muscarinic antagonist (GSK573719, 125mcg) combination therapy will be taken once daily for 4 weeks.
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 14 | 14
units on a scale | 3.9 (2.4) | 3.4 (2.3)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.090, t-test, 2 sided

2. Secondary Outcome: Exercise Endurance Time
Description: Duration of constant work rate cycle exercise at 75% of maximum
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 14 | 14
minutes | 7.82 (6.15) | 7.49 (4.99)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.680, t-test, 2 sided

3. Secondary Outcome: Inspiratory Capacity at Rest
Description: Measurements of pulmonary function included spirometry and body plethysmography. The resting inspiratory capacity (IC) values reported here are 90 minutes post-dose after 4 weeks of treatment.
Time Frame: 4 weeks
Population: 14 subjects completed both treatments for comparison.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 14 | 14
L | 2.27 (0.40) | 2.36 (0.86)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.197, t-test, 2 sided

4. Secondary Outcome: Ventilation at Isotime Exercise
Description: Ventilation was measured during constant work rate exercise tests. Isotime was defined as the highest exercise time in minutes common to both post-treatment tests.
Time Frame: 4 weeks
Population: 14 subjects completed both treatment arms for comparison.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 14 | 14
L/min | 44.9 (16.3) | 47.5 (18.4)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.006, t-test, 2 sided

5. Secondary Outcome: Intensity of "Unpleasantness of Breathing" at Isotime Exercise
Description: Intensity rating (modified 10-point Borg scale) measured at a standardized time (isotime) during constant work rate exercise tests. A rating of 0 represents no "unpleasantness of breathing" up to a maximum of 10. An improvement would be noted as a decrease in the Borg scale rating. Isotime was defined as the highest exercise time in minutes common to both post-treatment tests.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 14 | 14
units on a scale | 4.0 (2.5) | 3.3 (2.3)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.044, t-test, 2 sided

6. Secondary Outcome: Inspiratory Capacity at Isotime Exercise
Description: Measurements of inspiratory capacity (IC) were conducted during constant work rate exercise tests. Isotime was defined as the highest time in minutes completed in both post-treatment tests.
Time Frame: 4 weeks
Population: 14 subjects completed both treatment arms for comparison.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 14 | 14
L | 1.99 (0.56) | 2.02 (0.59)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.573, t-test, 2 sided

7. Secondary Outcome: Diaphragm Electromyogram (EMGdi) at Isotime Exercise
Description: EMGdi was measured during constant work rate exercise tests via a multipair-electrode esophageal catheter. EMGdi expressed as a percentage of its maximum is used as an index of inspiratory neural drive. Isotime was defined as the highest exercise time in minutes common to both post-treatment tests.
Time Frame: 4 weeks
Population: Although 14 subjects completed both treatment arms, only 9 subjects had complete measurements of EMGdi and respiratory pressures.
Measure: Mean (Standard Deviation); unit: percentage of maximum EMGdi
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 9 | 9
percentage of maximum EMGdi | 53.4 (17.4) | 53.5 (13.5)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.960, t-test, 2 sided

8. Secondary Outcome: Tidal Esophageal Pressure (Pes) Swings at Isotime Exercise
Description: Tidal esophageal pressure (Pes) swings were measured via an esophageal balloon catheter during constant work rate exercise tests. Tidal Pes expressed relative to maximum is an index of respiratory effort. Isotime was defined as the highest exercise time in minutes common to both post-treatment tests.
Time Frame: 4 weeks
Population: Although 14 subjects completed both treatment arms for comparison, only 9 subjects also had complete measurements of EMGdi and respiratory pressures.
Measure: Mean (Standard Deviation); unit: percentage of maximum Pes
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 9 | 9
percentage of maximum Pes | 28 (17) | 28 (20)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.944, t-test, 2 sided

9. Secondary Outcome: Mean Expiratory Flow at Isotime Exercise
Description: Mean expiratory flow was measured during constant work rate exercise tests. Isotime was defined as the highest exercise time in minutes common to both post-treatment tests.
Time Frame: 4 weeks
Population: 14 subjects completed both treatment arms for comparison.
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 14 | 14
L/s | 2.19 (0.80) | 2.34 (0.92)
Statistical Analysis 1: Comparison: LAMA vs LABA/LAMA Combination; A paired t-test using a 2-sided test of significance was used to compare values after LAMA versus LABA/LAMA treatment; Test type: Superiority; p = 0.028, t-test, 2 sided

10. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Measurements of pulmonary function included spirometry and body plethysmography. Values reported are 90 minutes post-dose after 4 weeks of treatment.
Time Frame: 4 weeks
Population: 14 subjects completed both treatments for comparison.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | LAMA | LABA/LAMA Combination
Number analyzed (Participants) | 14 | 14
L | 1.56 (0.40) | 1.72 (0.46)

ADVERSE EVENTS:
Time Frame: Over the duration of the study (approximately 12 weeks).
Groups:
- LAMA Arm: The 4-week treatment period with once daily inhaled umeclidinium (125 mcg).
- LABA/LAMA Arm: The 4-week treatment period with once daily inhaled fixed-dose combination of umeclidinium (125 mcg) and vilanterol (25 mcg).
- Washout Period: There was a 2 week washout period between the two treatment arms.
Arm/Group | LAMA Arm | LABA/LAMA Arm | Washout Period
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/17 | 0/17 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LAMA Arm (N=17) | LABA/LAMA Arm (N=17) | Washout Period (N=17)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — An exacerbation of COPD requiring treatment (oral steroids and/or antibiotic).
Pancreatitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No